CLINICAL TRIAL: NCT00405613
Title: Aspirin Use and Postoperative Bleeding From Dental Extractions in a Healthy Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSF-201090
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2006-11

CONDITIONS: Bleeding Complication
Keywords: Aspirin; Bleeding; Clinical Trial; Dental Extraction
MeSH Terms: conditions — Hemorrhage | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
The purpose of this study is to determine if aspirin is associated with bleeding complications following a single tooth extraction

DETAILED DESCRIPTION:
Aspirin is a common chronically administered preventive treatment for cardiovascular disease, but is often discontinued prior to invasive dental procedures because of concern of bleeding complications. As the goal of aspirin is often to prevent MI and stroke, the risk of these CVD outcomes with discontinuation of aspirin must be weighed against the perceived adverse event of bleeding during or following an invasive dental procedure with continuation of aspirin. The current study is a randomized controlled trial evaluating bleeding complications of aspirin vs. placebo in healthy patients schedule for a single tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Require a simple tooth extraction

Exclusion Criteria:

* Use of previous aspirin or NSAID

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-05; Study Completion 2005-12

PRIMARY OUTCOMES:
Oral bleeding time

SECONDARY OUTCOMES:
Report of bleeding at phone follow-up at 3-7 (first follow-up) and 40-55 hours (second follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Brennan, DDS,MHS, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States